CLINICAL TRIAL: NCT05852470
Title: PMCF (Post Market Clinical Follow-up) Evaluation of Clareon Vivity/Vivity Toric
Brief Title: Evaluation of Clareon Vivity/Vivity Toric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ILE632-C002
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Aphakia
Keywords: Cataract; Intraocular lens
MeSH Terms: conditions — Aphakia; Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors will be masked to the IOLs that have been previously implanted in the subject until the end of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Clareon Vivity/Vivity Toric (Experimental): Previous implantation in both eyes with Clareon Vivity/Vivity Toric Extended Vision IOL (intraocular lens), with previous implantation defined as 90-180 days post second eye implantation
  Interventions: Device: Clareon Vivity/Vivity Toric Extended Vision IOL
- Clareon Monofocal/Clareon Toric (Active Comparator): Previous implantation in both eyes with Clareon Monofocal/Clareon Toric IOL (intraocular lens), with previous implantation defined as 90-180 days post second eye implantation
  Interventions: Device: Clareon Monofocal/Clareon Toric IOL

INTERVENTIONS:
Device: Clareon Vivity/Vivity Toric Extended Vision IOL — Extended vision intraocular lens implanted in the capsular bag of the eye during cataract surgery. IOLs are intended for long term use over the lifetime of the cataract patient.
  Other Names: Models CNWET0, CNWET3, CNWET4, CNWET5, CNWET6, CCWET0, CCWET3, CCWET4, CCWET5, CCWET6; Clareon Vivity™ Extended Vision Hydrophobic IOL; Clareon Vivity™ Toric Extended Vision Hydrophobic IOL
  Arms: Clareon Vivity/Vivity Toric
Device: Clareon Monofocal/Clareon Toric IOL — Single vision intraocular lens implanted in the capsular bag of the eye during cataract surgery. IOLs are intended for long term use over the lifetime of the cataract patient.
  Other Names: SY60WF, CNW0T3, CNW0T4, CNW0T5, CNW0T6, CC60WF, CCW0T3, CCW0T4, CCW0T5, CCW0T6, Clareon with AutonoMe (CCA0T0, CNA0T0); Clareon™ Aspheric Hydrophobic Acrylic IOL; Clareon™ Toric Aspheric Hydrophobic Acrylic IOL
  Arms: Clareon Monofocal/Clareon Toric

SUMMARY:
This study seeks to generate clinical data from subjects previously implanted with the Clareon Vivity/Vivity Toric Intraocular Lenses (IOLs) or Clareon Monofocal/Clareon Toric IOLs. This study will assess key performance endpoints to support clinical benefits statements with model-specific data.

DETAILED DESCRIPTION:
Both eyes of a subject must qualify for enrollment into this study. A total of 2 scheduled visits are planned. The visits include a Screening visit (Visit 0) and a visit after screening (Visit 1). The subject must be 90-180 days post second eye implant at the time of Visit 1. Visit 1 should occur 1 to 14 days after Visit 0. Subject participation is expected to last approximately 2 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Understand and sign an approved Informed Consent form
* Previously implanted in both eyes with Clareon Vivity/Clareon Vivity Toric or Clareon Monofocal/Clareon Toric IOLs for at least 3 months and up to 6 months (90 to 180 days) after second eye implant.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* History of clinically significant ocular co-morbidities that would affect surgical outcomes based on investigator expert medical opinion.
* Subjects who were targeted to monovision defined as ≥ 1.50 Diopter (D) of anisometropia.
* Clinically significant PCO (posterior capsule opacification) affecting vision.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Surgical CRD, Study Director — Alcon Research, LLC
Locations (7):
- United States (7):
  - Wolstan Goldberg Eye Associates, Torrance, California
  - Eye Center of Northern Colorado, PC, Fort Collins, Colorado
  - Grosinger, Spigelman & Grey Eye Surgeons, P.C., Bloomfield Hills, Michigan
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Eye Care Specialists, Kingston, Pennsylvania
  - Carolina Eyecare Physicians LLC, Mt. Pleasant, South Carolina
  - Vance Thompson Vision, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 7 investigative sites located in the United States.
Pre-assignment Details: Of the 155 enrolled, 5 participants were exited as screen failures. This reporting group includes all eligible subjects (150).
Period: Overall Study
Arm/Group | Clareon Vivity/Vivity Toric | Clareon Monofocal/Clareon Toric
Started | 73 | 77
Full Analysis Set | 73 | 76
Completed | 73 | 76
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All subjects/eyes bilaterally implanted with the test or comparator IOL
Groups:
- Total: Total of all reporting groups
Arm/Group | Clareon Vivity/Vivity Toric | Clareon Monofocal/Clareon Toric | Total
Number analyzed (Participants) | 73 | 76 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (8.92) | 71.5 (6.97) | 70.0 (8.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 46 | 88
  Male | 31 | 30 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 73 | 75 | 148
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 68 | 63 | 131
  Black or African American | 2 | 7 | 9
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 73 | 76 | 149

OUTCOME MEASURES:

1. Primary Outcome: Mean Binocular Photopic Best Corrected Distance Visual Acuity (BCDVA) at 3 to 6 Months (90 to 180 Days) Postoperatively After Second Eye Implant
Description: Visual acuity (VA) was assessed with best refractive correction in place under photopic (well-lit) conditions at a distance of 4 meters (m) using a visual acuity chart. VA was measured in logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity, with a lower logMAR value indicating better visual acuity. This was a subject-based assessment. Both eyes were assessed together. This is a co-primary endpoint.
Time Frame: Visit 1 (Day 1-14 post Screening Visit, coinciding with Day 90-180 post second eye implantation)
Population: FAS. Note: One subject in the Clareon Monofocal/Clareon Toric arm discontinued after Visit 0; thus, the data from this subject at this visit is not included.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Clareon Vivity/Vivity Toric | Clareon Monofocal/Clareon Toric
Number analyzed (Participants) | 73 | 75
logMAR | -0.028 (0.1165) | -0.062 (0.0847)
Statistical Analysis 1: Comparison: Clareon Vivity/Vivity Toric vs Clareon Monofocal/Clareon Toric; Test type: Non-Inferiority — Non-inferiority margin = 0.1 logMAR; Since a non-inferiority hypothesis is being tested, a p-value is not applicable. Confidence limit is being reported and compared to the non-inferiority margin; Difference in Means = 0.034, 95% CI 2-sided [0.001 to 0.067], Standard Error of Mean 0.0167 — Parameter Dispersion Type is Standard Error of the Difference in Means. Difference = Vivity/Vivity Toric Extended Vision IOL minus Clareon/Clareon Toric Monofocal IOL

2. Primary Outcome: Mean Binocular Photopic Distance Corrected Intermediate Visual Acuity (DCIVA) at 3 to 6 Months (90 to 180 Days) Postoperatively After Second Eye Implant
Description: Visual acuity (VA) was assessed with distance correction in place (plus or minus power) under photopic (well-lit) conditions at a distance of 66 centimeters (cm) from the spectacle plane using a visual acuity chart. VA was measured in logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity, with a lower logMAR value indicating better visual acuity. This was a subject-based assessment. Both eyes were assessed together. This is a co-primary endpoint.
Time Frame: Visit 1 (Day 1-14 post Screening Visit, coinciding with Day 90-180 post second eye implantation)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Clareon Vivity/Vivity Toric | Clareon Monofocal/Clareon Toric
Number analyzed (Participants) | 73 | 75
logMAR | 0.035 (0.0788) | 0.126 (0.1033)
Statistical Analysis 1: Comparison: Clareon Vivity/Vivity Toric vs Clareon Monofocal/Clareon Toric; Test type: Superiority; p < .001, t-test, 1 sided; Difference in Means = -0.091, 95% CI 2-sided [-0.120 to -0.061], Standard Error of Mean 0.0151; Parameter Dispersion Type is Standard Error of the Difference in Means. Difference = Vivity/Vivity Toric Extended Vision IOL minus Clareon/Clareon Toric Monofocal IOL

3. Secondary Outcome: Mean Binocular Photopic Distance Corrected Near Visual Acuity (DCNVA) at 3 to 6 Months (90 to 180 Days) Postoperatively After Second Eye Implant
Description: Visual acuity (VA) was assessed with distance correction in place (plus or minus power) under photopic (well-lit) conditions at a distance of 40 centimeters (cm) from the spectacle plane using a visual acuity chart. VA was measured in logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity, with a lower logMAR value indicating better visual acuity. This was a subject-based assessment. Both eyes were assessed together.
Time Frame: Visit 1 (Day 1-14 post Screening Visit, coinciding with Day 90-180 post second eye implantation)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Clareon Vivity/Vivity Toric | Clareon Monofocal/Clareon Toric
Number analyzed (Participants) | 73 | 75
logMAR | 0.205 (0.1008) | 0.334 (0.1410)
Statistical Analysis 1: Comparison: Clareon Vivity/Vivity Toric vs Clareon Monofocal/Clareon Toric; Test type: Superiority; p < .001, t-test, 1 sided; Difference in Means = -0.129, 95% CI 2-sided [-0.169 to -0.089], Standard Error of Mean 0.0202 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Subjects Who Respond "Never" to Question 1 of the Intraocular Lens Satisfaction (IOLSAT) Questionnaire at 3 to 6 Months (90 to 180 Days) Postoperatively After Second Eye Implant
Description: The IOLSAT is a patient-reported outcomes questionnaire. Subjects were asked, "Overall, in the past 7 days, how often did you need to wear eyeglasses to see?" The percentage was calculated as (# of subjects responding "Never") divided by (# of subjects with bilateral implantation and concordant, non-missing data) times 100. A higher percentage is a better outcome.
Time Frame: Visit 1 (Day 1-14 post Screening Visit, coinciding with Day 90-180 post second eye implantation)
Population: FAS with requisite data at visit. Note: One subject in the Clareon Monofocal/Clareon Toric arm discontinued after Visit 0; thus, the data from this subject at this visit is not included.
Measure: Number; unit: percentage of participants
Arm/Group | Clareon Vivity/Vivity Toric | Clareon Monofocal/Clareon Toric
Number analyzed (Participants) | 70 | 73
percentage of participants | 21.4 | 4.1
Statistical Analysis 1: Comparison: Clareon Vivity/Vivity Toric vs Clareon Monofocal/Clareon Toric; Test type: Superiority; Miettinen-Nurminen — The lower boundary of the confidence interval is reported instead of a p-value; Difference in Percentages = 17.32, 90% CI 2-sided [lower limit 8.66] (Upper limit is not applicable for testing.) — Difference = Vivity/Vivity Toric Extended Vision IOL minus Clareon/Clareon Toric Monofocal IOL

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent until study exit. The total expected duration of participation for each subject was approximately 14 days.
Description: AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is included with unit of "eyes." The Other (Not Including Serious) Adverse Event table reports only the AEs that occurred above a 5% threshold in one or more reporting group. This analysis population includes all subjects/eyes bilaterally implanted with the test or comparator IOL.
Groups:
- Clareon Vivity/Vivity Toric - First Eye (Ocular): All first study eyes previously implanted with Clareon Vivity/Vivity Toric IOL
- Clareon Vivity/Vivity Toric - Second Eye (Ocular): All second study eyes previously implanted with Clareon Vivity/Vivity Toric IOL
- Clareon Vivity/Vivity Toric - Systemic: All subjects implanted with Clareon Vivity/Vivity Toric IOL
- Clareon Monofocal/Clareon Toric - First Eye (Ocular): All first study eyes previously implanted with Clareon Monofocal/Clareon Toric IOL
- Clareon Monofocal/Clareon Toric - Second Eye (Ocular): All second study eyes previously implanted with Clareon Monofocal/Clareon Toric IOL
- Clareon Monofocal/Clareon Toric - Systemic (Subject): All subjects implanted with Clareon Monofocal/Clareon Toric IOL
Arm/Group | Clareon Vivity/Vivity Toric - First Eye (Ocular) | Clareon Vivity/Vivity Toric - Second Eye (Ocular) | Clareon Vivity/Vivity Toric - Systemic | Clareon Monofocal/Clareon Toric - First Eye (Ocular) | Clareon Monofocal/Clareon Toric - Second Eye (Ocular) | Clareon Monofocal/Clareon Toric - Systemic (Subject)
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/73 | 0/73 | 0/76 | 0/76 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/73 | 0/73 | 0/76 | 0/76 | 0/76
Other Adverse Events (participants affected / at risk) | 0/73 | 0/73 | 0/73 | 0/76 | 0/76 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT05852470/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT05852470/SAP_001.pdf